CLINICAL TRIAL: NCT03469609
Title: A Randomized Multicenter Open-label Controlled Trial to Show That Mucous Fistula Refeeding Reduces the Time From Enterostomy Closure to Full Enteral Feeds (MUCous FIstula REfeeding ("MUC-FIRE") Trial)
Brief Title: Mucous Fistula Refeeding Reduces the Time From Enterostomy Closure to Full Enteral Feeds ("MUC-FIRE" Trial)
Acronym: MUC-FIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: German Research Foundation (Other); Hannover Medical School (Other)
Responsible Party: Principal Investigator, Martin Lacher, Prof. Dr. med., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUC-FIRE
Record Dates: First submitted 2018-02-28; First posted 2018-03-19 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Enterostomy
Keywords: infants; necrotizing enterocolitis (NEC); focal intestinal perforation (FIP); enterostomy creation; bowel reanastomosis; enteral feeding; caloric intake; parenteral nutrition; complication rate; reduction of hospital expenses; length of hospital stay; refeeding
MeSH Terms: conditions — Enterocolitis, Necrotizing; Hyperphagia

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, randomized, parallel group, controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative mucous fistula refeeding (Experimental): Perioperative mucous fistula refeeding between enterostomy creation and enterostomy closure
  Interventions: Other: mucous fistula refeeding
- No mucous fistula refeeding (No Intervention): No perioperative mucous fistula refeeding

INTERVENTIONS:
Other: mucous fistula refeeding — Transfer of infants' own stool
  Arms: Perioperative mucous fistula refeeding

SUMMARY:
The primary objective of this study is to demonstrate that mucous fistula refeeding between enterostomy creation and enterostomy closure reduces the time to full enteral feeds after enterostomy closure compared to standard of care.

DETAILED DESCRIPTION:
Enterostomies in children may be created for different reasons. During the presence of an enterostomy the regular stool transfer is interrupted as the distal part of the bowel (the part following the enterostomy) does not participate in the circulation of stool. Therefore it does not contribute to the resorption of enteral contents. As a consequence these children need additional parenteral nutrition. Due to the negative side-effects of parenteral nutrition all patients should return to enteral nutrition as soon as possible. Consequently, many pediatric surgical centers worldwide routinely perform mucous fistula refeeding (MFR) into the former unused bowel after enterostomy creation because case reports and retrospective analyses show low complication rates and faster postoperative weight gain. Several providers, however, shy away from this approach because to date there is still no high quality evidence for the benefit of this Treatment.The aim of this study is to assess the effects of mucous fistula refeeding in a randomized, prospective trial. We hypothesize that MFR between enterostomy creation and enterostomy closure reduces the time to full enteral feeds after enterostomy closure compared to the group without refilling. Moreover, the side effects of parenteral nutrition may be reduced and the postoperative hospital care of infants undergoing ostomy closure shortened.

ELIGIBILITY:
Inclusion Criteria:

1. Infants < 366 days,
2. Ileostomy / Jejunostomy,
3. double loop enterostomies and split enterostomies (with mucous fistula)
4. Signed written informed consent obtained by parents/legal guardians and willingness of parents/legal guardians to comply with treatment and follow-up procedures of their child

Exclusion Criteria:

1. resection of ileocecal valve,
2. colostomy,
3. small bowel atresia,
4. multiple ostomies (more than just an enterostomy and a mucous fistula),
5. chromosomal abnormalities (if known at the time of randomization),
6. Hirschsprung's disease,
7. participation in another drug-intervention study
8. Intestinal perforation due to a hemodynamic heart defect

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Time to full enteral feeds (hours) | week 4 to week 12 daily
  Time to full feeds (hours), defined as time to actual enteral intake of the age-dependent caloric requirements per day (defined as 90 or 120kcal/kg/24h) for at least 24 hours and a concomitant reduction of parenteral fluids to <20ml/kg/24h.
  1. The nutrition aim is 120 kcal/kg/24h for premature infants with a birth weight < 1000g or premature infants with a birth weight ≥ 1000g and mother's gestation week at birth before 37+0.
  2. The nutrition aim is 90 kcal/kg/24h for born mature infants, mother's gestation week at birth at least 37+0.

SECONDARY OUTCOMES:
Time to first bowel movement | Week 4 to week 12 daily
  Cleaning and changing of infants diapers will be performed according to a fixed schedule in order to uniformly document the time to first bowel movement
Thriving | Week 1 to week 12 daily; follow-up (month 3, 6, 12)
  Measurement of body weight
Z-Score (standard deviation score) | Week 1 to week 12 daily, follow-up (month 3, 6, 12)
  Measurement of weight [weight for age, World Health Organization (WHO)]
Number of days of postoperative total parenteral nutrition (TPN) | Week 2 to week 12 daily, follow-up (month 3, 6, 12)
  Calculation of days of postoperative TPN starts on the day of operation and ends on the day of full enteral nutrition
Laboratory parameter indicating cholestasis | Week 1 to week 12 daily, follow-up (month 3)
  Measurement of conjugated Bilirubin (µmol/l)
Assessment of adverse events (AEs) | Week 1 to week 12 daily, follow-up (month 3, 6, 12)
  Adverse events will be collected by the investigator either based on the information provided spontaneously by the parents of patient or evaluated by non-suggestive questions.
Assessment of serious adverse events (SAEs) | Week 1 to week 12 daily, follow-up (month 3, 6, 12)
  Adverse events will be collected by the investigator either based on the information provided spontaneously by the parents of patient or evaluated by non-suggestive questions.
Postoperative weight gain (g/d) | week 4 to week 12
  Weight gain during the subsequent 5 days after reaching the primary endpoint following enterostomy closure
Central venous line (CVL) | Week 1 to week 12
  duration (days) and number of CVL infections (definition of infection: Neo-Kiss Guidelines)
hospitalisation | week 1 to week 12
  Length of hospital stay (days)
jump in caliber | week 5
  Estimated ratio of the diameter of the two bowel loops which are anastomosed.
Sodium resorption | Week 1 to week 12 daily, follow-up (month 3)
  Sodium in Urine (mmol/l)
Status of liver enzymes | Week 1 to week 12 daily, follow-up (month 3)
  Gamma-Glutamyltransferase (GGT) , Alanine-Aminotransferase (ALT) , Aspartate-Aminotransferase (AST) (µkat/l)
Laboratory parameters | Week 1 to week 12 daily, follow-up (month 3)
  Haemoglobin (g/dl)
Time to full volume intake per day (in hours) | week 4 to week 12 daily
  Time to full age-dependent volume intake per day (defined as 150ml/kg/24h for premature infants and 120ml/kg/24h for mature born infants as well as corrected mature infants) (in hours).
  1. The volume aim is 150 ml/kg/24h for premature infants with a birth weight < 1000g or premature infants with a birth weight ≥ 1000g and mother's gestation week at birth before 37+0.
  2. The volume aim is 120 ml/kg/24h for born mature infants, mother's gestation week at birth at least 37+0.

CONTACTS AND LOCATIONS:
Overall Officials: Omid Madadi-Sanjani, Dr. med., Principal Investigator — Hannover Medical School, Department of Pediatric Surgery; Martin Lacher, Prof. Dr., Principal Investigator — University of Leipzig, Department of Pediatric Surgery
Locations (16):
- Austria (2):
  - Universitätsklinik für Kinder- und Jugendchirurgie, Graz
  - Universitätsklinik für Kinder- und Jugendheilkunde, Vienna
- Germany (12):
  - Universitätsklinik für Kinder- und Jugendmedizin Tübingen, Tübingen, Baden-Wurttemberg
  - Städtisches Klinikum München GmbH/ Klinikum Schwabing, München, Bavaria
  - Zentrum der Chirurgie, Klinik für Kinderchirurgie, Frankfurt am Main, Hesse
  - Auf der Bult, Kinder- und Jugendkrankenhaus, Kinderchirurgie und Kinderurologie, Hanover, Lower Saxony
  - Hannover Medical School, Clinic for Pediatric Surgery, Hanover, Lower Saxony
  - Marien Hospital Witten, Ruhr-University Bochum, Department of Pediatric Surgery, Witten, North Rhine-Westphalia
  - Universitätsmedizin Mainz, Klinik und Poliklinik für Kinderchirurgie, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Kinderchirurgie, Dresden, Saxony
  - University of Leipzig, Leipzig, Saxony
  - University Hospital Augsburg, Clinic for Pediatric Surgery, Augsburg
  - Hamburg [University Hospital Hamburg Eppendorf/UKE & Altonaer Kinderkrankenhaus/AKK], Hamburg
  - University Hospital Marburg, Clinic for Pediatric Surgery, Marburg
- Netherlands (2):
  - Amsterdam University Medical Centers, Amsterdam
  - Erasmus University Medical Center Rotterdam, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grosshennig A, Wiesner S, Hellfritsch J, Thome U, Knupfer M, Peter C, Metzelder M, Binder C, Wanz U, Flucher C, Brands BO, Mollweide A, Ludwikowski B, Koluch A, Scherer S, Gille C, Theilen TM, Rochwalsky U, Karpinski C, Schulze A, Schuster T, Weber F, Seitz G, Gesche J, Nissen M, Jager M, Koch A, Ure B, Madadi-Sanjani O, Lacher M. MUC-FIRE: Study protocol for a randomized multicenter open-label controlled trial to show that MUCous FIstula REfeeding reduces the time from enterostomy closure to full enteral feeds. Contemp Clin Trials Commun. 2023 Feb 20;32:101096. doi: 10.1016/j.conctc.2023.101096. eCollection 2023 Apr. PMID 36875554

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT03469609/Prot_SAP_004.pdf